CLINICAL TRIAL: NCT04006795
Title: A Photo-irritation and Photo-sensitisation Study in Healthy Subjects for Three Developmental Cosmetic Facial Products
Brief Title: A Photoxicity and Photoallergy Study of a Developmental Face Cream, Serum and Lotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 212378
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Skin Care
Keywords: Skin Care, Cosmetic Facial Product
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Developmental Serum (Experimental): All participants in induction phase will be topically applied 2 semi-occlusive patch (Monday) containing developmental serum (0.02milliliters per centimeter square[mL/cm^2] in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, developmental serum will be re-applied and 1 of the 2 sites will be irradiated with 2.5 Joules per centimeters square(J/cm^2) ultraviolet(UV) A radiation,then with 0.3 minimal erythemal doses(MEDs) of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants will be applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site will be irradiated (same as induction phase). Assessment will be after 24, 48 and 72 hours of irradiation
  Interventions: Other: Serum
- Developmental Lotion (Experimental): All participants in induction phase will be topically applied 2 semi-occlusive patch (Monday) containing developmental lotion (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, developmental lotion will be re-applied and 1 of the 2 sites will be irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants will be applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site will be irradiated (same as induction phase). Assessment will be after 24, 48 and 72 hours of irradiation
  Interventions: Other: Lotion
- Developmental Cream (Experimental): All participants in induction phase will be topically applied 2 semi-occlusive patch (Monday) containing developmental cream (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, developmental cream will be re-applied and 1 of the 2 sites will be irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants will be applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site will be irradiated (same as induction phase). Assessment will be after 24, 48 and 72 hours of irradiation
  Interventions: Other: Cream
- Negative Control (Placebo Comparator): All participants in induction phase will be topically applied 2 semi-occlusive patch (Monday) containing 0.9 percent normal saline (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, normal saline will be re-applied and 1 of the 2 sites will be irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants will be applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site will be irradiated (same as induction phase). Assessment will be after 24, 48 and 72 hours of irradiation
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Serum — Participants will be topically applied adhesive patch containing developmental serum
  Arms: Developmental Serum
Other: Lotion — Participants will be topically applied adhesive patch containing developmental lotion
  Arms: Developmental Lotion
Other: Cream — Participants will be topically applied adhesive patch containing developmental cream
  Arms: Developmental Cream
Other: Normal Saline — Participants will be topically applied adhesive patch containing normal saline
  Arms: Negative Control

SUMMARY:
The purpose of this study is to demonstrate the absence of sensitisation and irritation potential of a product when applied to the skin and exposed to ultraviolet (UV) radiation. Photo-sensitisation potential will primarily be evaluated through a subsequent semi-occluded application and UV exposure (challenge phase) after a 2-week rest period. Photo-irritation potential will primarily be evaluated through the repeated occluded application and UV exposure of the study products over 3 weeks (induction phase).

DETAILED DESCRIPTION:
A single-center, randomised, evaluator (single) blind study in healthy adult participants aged 18 to 65 years with no dermatological disorders to evaluate the cutaneous photo- irritation and photo-sensitisation potential of three cosmetic facial skincare products. During Screening (Visit 1), the participants will sign an informed consent, will undergo dermatological assessment to ensure they have no dermatoses on their dorsum that might impact their safety, Fitzpatrick Phototype of II to IV and colorimetry analysis of their skin type using the Individual Typology Angle, which will be used to estimate minimal erythemal dose (MED). At Visit 2, the eligible participants will undergo MED irradiation where the participant will be administered a series of 6 controlled doses of UV radiation. At Visit 3, the participants will undergo MED determination, where a trained evaluator will evaluate the exposed skin to determine the lowest dose of UV radiation required to induce uniform, unambiguous erythema for signs of visible erythema. Further, the study will progress in 3-phases: Induction phase, Rest Phase and Challenge Phase. The Induction phase (3 weeks: Visit 4 to Visit 18); at visit 4, the area for applying 2 consecutive patches will be designated between the scapula and waistline. A controlled amount (0.02 mL/cm^2) of each study product will be randomly assigned within the patch system of each participant into the appropriate separate cell (3 cells for each of the test products and 1 cell for the saline solution). Every Monday, patch sites will be evaluated, 2 patches will be applied, post 24 hours (Tuesday) the patches will be removed, patch sites can be cleaned, patch sites will be evaluated, test products/ saline will be re-applied and 1 of the 2 sites will be irradiated with 2.5 Joules per centimetre square UVA radiation with a Schott UG11+WG335 filter (or equivalent) in place, and then with 0.3 MEDs of UVA+UVB radiation (filters UG11+WG320). The sites will be assessed immediately after irradiation and 24 hours post irradiation (Wednesday) and duplicate patches will be re-applied as applied on Monday. Same procedure will be repeated on Thursday as done on Tuesday and on Friday the patch sites will be evaluated. The same process will continue for 3 consecutive weeks. Then there will be 2 weeks of Rest phase; where there will be no product or patch applications. Rest phase is further followed by Challenge phase at week 6 (Visit 19 to Visit 23) where there will be a duplicate parallel series of product applications under semi-occlusive patches to 2 naïve areas on Monday. Post 24 hours (Tuesday) patches will be removed and 1 of the 2 sites will be irradiated similar as done in induction phase. The sites will be assessed immediately post irradiation and after 24 hours (Tuesday), 48 hours (Wednesday) and 72 hours (Thursday) of irradiation. At visit 23, after the challenge phase the final assessments will be performed by the dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon dermal examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant with Fitzpatrick phototype II to IV.
* A participant with healthy, intact skin at the proposed test area dorsum (below the shoulder, above the waist), as evaluated by a dermatologist, to ensure participant is free of clinically relevant dermatological conditions.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies involving investigational product(s) within 30 Days prior to study entry and/or during study participation.
* A participant who has participated in other studies including non-medicinal, cosmetic studies within 7 Days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant (self-reported).
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials/product (or closely related compounds) or any of their stated ingredients, to hypoallergenic tape, or to the cotton patches.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the Lifestyle Considerations; a) applying other product to test site, using cosmetics, b) changing dietary habits, c) getting patch test site wet, d) removing the patch, e) wearing tight or restrictive clothing that can remove patch, f) engaging in activities that result in excessive sweating, and g) intentional exposure to artificial ultraviolet light or cosmetic procedures.
* A participant with current or recent (within last 6 months before the start of the study) history of atopic lesions and/or eczema, psoriasis or skin cancer.
* A participant with a history of allergic reactions to topical-use products, cosmetics or medications or their ingredients.
* A participant with any history of significant diseases or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* A participant considered immune-compromised.
* A participant with active dermatosis (local or disseminated) that might interfere with the results of the study.
* A Participant with history of diseases aggravated or triggered by ultraviolet radiation.
* A participant currently using any medication, which in the opinion of the investigator, may affect the evaluation of the investigational product, or place the participant at undue risk (e.g. any photosensitising medication such as tetracycline, thiazides, fluoroquinolones, etc.) within one month prior to inclusion.
* A participant who has used any of the following topical or systemic medications up to two weeks before the screening visit: immuno-suppressants, antihistamines, nonsteroidal anti-inflammatory drugs (NSAIDS), and particular aspirin (>200mg/d), within two weeks prior to inclusion and/or corticosteroids.
* A participant who has used oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* A participant who has been vaccinated up to 1 month before the screening visit or is intending to receive a vaccination during their participation in the study.
* Currently receiving allergy injections or received an allergy injection within 7 days prior to Visit 1 or expects to begin injections during study participation.
* A participant with any skin marks on the back that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles, open sores, pimples, or cysts).
* A participant that intends bathing (in the sea or a pool), using a sauna, or partaking in water sports, or activities that lead to intense sweating for the duration of the study.
* A participant who has used a transcutaneous electrical nerve stimulation (TENS) machine 1 day before the screening visit or intends to use a TENS machine at any point during the study.
* A participant with history of sensitisation in a previous patch study.
* A participant with history of abnormal reaction to sun exposure.
* A participant who had intense sunlight exposure or sun tanning sessions up to 30 days before the screening evaluation.
* A participant with recent history (within the last 5 years) of alcohol or other substance abuse.
* A participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Brazil.
Pre-assignment Details: A total of 61 participants were screened, of which 40 participants were enrolled and 37 participants were randomized, 3 enrolled participants were not randomized as they missed scheduled site visits. All 37 randomized participants completed the study.
Groups:
- Overall Participants: All participants in 3 week induction phase topically applied 2 semiocclusive patch (0.02milliliters per centimeter square[mL/cm^2])on Monday, containing developmental serum,lotion,cream,negative control(Sodium Chloride[NaCl:0.9percent{%}])at 2sites on dorsum for 24hours.Post patch removal(Tuesday)sites cleaned,developmental serum reapplied,1site irradiated with 2.5Joules per centimeters square(J/cm^2)ultraviolet(UV)A radiation,then with 0.3minimal erythemal doses(MEDs)of UVA+UVB radiation.Duplicate test site not exposed to UVradiation.24hours post irradiation(Wednesday),sites assessed,duplicate patches applied as on Monday.Irradiation on Thursday similar to Tuesday,assessment post 24hour on Friday.Participants then entered 2week rest phase(no product or patch applications) followed by challenge phase where all participants applied 2semiocclusive patches at 2naive sites for 24hours,1site irradiated(like induction phase).Assessment done after 24,48,72 hours of irradiation till Day40.
Period: Induction Phase
Arm/Group | Overall Participants
Started | 37
Completed | 37
Not Completed | 0
Period: Rest Phase
Arm/Group | Overall Participants
Started | 37
Completed | 37
Not Completed | 0
Period: Challenge Phase
Arm/Group | Overall Participants
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all randomized participants who received at least 1 dose of any study product.
Groups:
- Overall Participants: All participants in 3 week induction phase topically applied 2 semiocclusive patch (0.02 mL/cm^2)on Monday, containing developmental serum,lotion,cream,negative control(NaCl: 0.9 %)at 2 sites on dorsum for 24 hours.Post patch removal (Tuesday) sites cleaned,developmental serum reapplied,1 site irradiated with 2.5 J/cm^2 UVA radiation,then with 0.3 MEDs of UVA+UVB radiation.Duplicate test site not exposed to UVradiation. 24hours post irradiation(Wednesday),sites assessed,duplicate patches applied as on Monday.Irradiation on Thursday similar to Tuesday,assessment post 24 hour on Friday.Participants then entered 2 week rest phase(no product or patch applications) followed by challenge phase where all participants applied 2 semiocclusive patches at 2 naive sites for 24 hours, 1 site irradiated(like induction phase).Assessment done after 24,48,72 hours of irradiation till Day 40.
Arm/Group | Overall Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type Grading [Number; unit: Number of Participants] — Fitzpatrick scale was used to classify a participant's skin type by their response to sun exposure. This scale emphasizes on potentials for irritation, burns and hyperpigmentation, indicators for future product choices. This scale has six grading, where I refers to always burns easily; never tans, II refers to always burns easily; tans minimally, III refers to burns moderately; tans gradually, IV refers to burns minimally, always tans well, V refers to rarely burns, tans profusely and VI refers to never burns.
  Number of Participants
    Fitzpatrick Skin Type Grading | 37
    I - Pale white skin | 0
    II - White skin | 5
    III - Light brown skin | 20
    IV - Moderate brown skin | 12
    V - Dark brown skin | 0
    VI - Deeply pigmented dark brown to black skin | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Photo-initiated Potential Sensitization Reaction
Description: Scoring of patch test reactions was performed by blind evaluator as per International Contact Dermatitis Research Group (ICDRG) grading '- to +++',where '-':negative reaction;'?+':doubtful reaction(faint erythema only),'+':weak(non-vesicular) positive reaction(erythema, infiltration and possibly papules);'++':strong(vesicular) positive reaction (erythema,infiltration,papules,vesicles); '+++':extreme positive reaction (bullous reaction, intense erythema and infiltration, coalescing vesicles).Score range '- to +++' where '-' indicated no adverse reaction and '+++' indicated very strong adverse reaction.Any positive reaction ('+' or greater):considered potential sensitization(PS) upon dermatologist discretion and as potential photo-initiated if a)positive reaction occur at ultraviolet (UV) exposed site,b)occur at both UV and non-UV sites with maximum score at UV exposed site being higher than non-UV exposed site.Percentage of participants with photo-initiated PS were reported in numbers.
Time Frame: Day 40
Population: The Safety Population included all randomized participants who received at least 1 dose of any study product.
Measure: Number; unit: Participants
Groups:
- Developmental Serum: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental serum (0.02 mL/cm^2) in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites were cleaned, developmental serum was re-applied and 1 of the 2 sites were irradiated with 2.5 J/cm^2 UV A radiation,then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
- Developmental Lotion: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental lotion (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, developmental lotion was re-applied and 1 of the 2 sites were irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
- Developmental Cream: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental cream (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites were cleaned, developmental cream was re-applied and 1 of the 2 sites were irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
- Negative Control: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing 0.9 percent normal saline (0.02mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, normal saline was re-applied and 1 of the 2 sites was irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With a Photo-initiated Reaction (Score of '+' or Greater) Which is Not Considered Potential Sensitization Reaction
Description: Scoring of patch test reactions was performed by blind evaluator as per ICDRG grading '- to +++', where '-':negative reaction; '?+':doubtful reaction(faint erythema only),'+':weak(non-vesicular) positive reaction(erythema, infiltration and possibly papules);'++':strong(vesicular) positive reaction (erythema, infiltration, papules, vesicles);'+++':extreme positive reaction (bullous reaction, intense erythema and infiltration, coalescing vesicles).Score range '- to +++' where '-' indicated no adverse reaction and '+++' indicated very strong adverse reaction.Any positive reaction ('+' or greater) was classified as photo-initiated if a) a positive reaction occurs only at UV exposed site,b) occur at both UV and non-UV site with maximum score at UV exposed site being higher than maximum score at non-UV exposed site. Percentage of participants with any photo-initiated reaction (score of '+' or greater) without potential sensitisation were reported in form of numbers.
Time Frame: Day 40
Population: The Safety Population included all randomized participants who received at least 1 dose of any study product.
Measure: Number; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 37 | 37 | 37 | 37
Participants | 0 | 0 | 1 | 0

3. Secondary Outcome: Percentage of Participants With a Potential Sensitization Reaction Which is Not Considered Photo-initiated
Description: Scoring of patch test reactions was performed by blind evaluator as per ICDRG grading grading '- to +++', where '-':negative reaction; '?+':doubtful reaction(faint erythema only),'+':weak(non-vesicular) positive reaction(erythema, infiltration and possibly papules); '++':strong(vesicular) positive reaction (erythema, infiltration, papules and vesicles); '+++':extreme positive reaction (bullous reaction, intense erythema and infiltration, coalescing vesicles). Score range '- to +++' where '-' indicates no adverse reaction and '+++' indicates very strong adverse reaction.Any positive reaction (a score of '+' or greater) was considered as potential sensitization based upon dermatologist discretion and was further considered as non-photoinitiated if: a positive reaction occurs only at the non-UV exposed site. Percentage of participants with any non-photoinitiated potential sensitisation was reported in form of numbers.
Time Frame: Day 40
Population: The Safety Population included all randomized participants who received at least 1 dose of any study product.
Measure: Number; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With a Non-photoinitiated Reaction (Score of '+' or Greater) Which is Not Considered Potential Sensitization Reaction
Description: Scoring of patch test reactions was performed by blind evaluator as per ICDRG grading grading '- to +++', where '-':negative reaction; '?+':doubtful reaction(faint erythema only),'+':weak(non-vesicular) positive reaction(erythema, infiltration and possibly papules); '++':strong(vesicular) positive reaction (erythema, infiltration, papules and vesicles); '+++':extreme positive reaction (bullous reaction, intense erythema and infiltration, coalescing vesicles). Score range '- to +++' where '-' indicates no adverse reaction and '+++' indicates very strong adverse reaction.Any positive reaction (a score of '+' or greater) was considered as non-photoinitiated if: a positive reaction occurs only at the non-UV exposed site. Percentage of participants with non-photoinitiated reaction (score of '+' or greater) without potential sensitization was reported in form of numbers.
Time Frame: Day 40
Population: The Safety Population included all randomized participants who received at least 1 dose of any study product.
Measure: Number; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control
Number analyzed (Participants) | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 40
Description: The Safety Population included all randomized participants who received at least 1 dose of any study product. All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported.
Groups:
- Developmental Serum: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental serum (0.02 mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites were cleaned, developmental serum was re-applied and 1 of the 2 sites were irradiated with 2.5 J/cm^2 UV A radiation,then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
- Developmental Lotion: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental lotion (0.02 mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, developmental lotion was re-applied and 1 of the 2 sites were irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
- Developmental Cream: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing developmental cream (0.02 mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites were cleaned, developmental cream was re-applied and 1 of the 2 sites were irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites were assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40..
- Negative Control: All participants in induction phase were topically applied 2 semi-occlusive patch (Monday) containing 0.9 percent normal saline (0.02 mL/cm^2 in an individual cell of patch) at 2 sites on the dorsum for 24 hours, post patch removal(Tuesday), sites will be cleaned, normal saline was re-applied and 1 of the 2 sites was irradiated with 2.5J/cm^2 UVA radiation, then with 0.3 MEDs of UVA+UVB radiation. 24 hours post irradiation (Wednesday), sites will be assessed and duplicate patches applied as on Monday for 24 hours. Irradiation on Thursday similar to Tuesday and assessment post 24 hour irradiation on Friday. Same process repeated for 3 weeks. In challenge phase all participants were applied 2 semi-occlusive patches at 2 naive sites for 24 hours, post which 1 site was irradiated (same as induction phase). Assessment was done after 24, 48 and 72 hours of irradiation till day 40.
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Negative Control | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 8/37 | 8/37 | 8/37 | 8/37 | 8/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Developmental Serum (N=37) | Developmental Lotion (N=37) | Developmental Cream (N=37) | Negative Control (N=37) | Overall Participants (N=37)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Herpes virus infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT04006795/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT04006795/SAP_001.pdf